CLINICAL TRIAL: NCT00923975
Title: Evaluation of Avatar Web Reports
Brief Title: Evaluation of DIDGET TM World Reports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2009-08
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2010-10-08 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the Software (Other): Young adults, parents/guardians of young people under age 18, and healthcare professionals who work with this population would be intended users of the data management program. The DIDGET World Reports software is used to upload blood glucose results from the DIDGET Blood Glucose Monitoring System so that intended users can identify patterns in their diabetes management.
  Interventions: Device: DIDGET World Web Community Reports

INTERVENTIONS:
Device: DIDGET World Web Community Reports — During the study subjects performed specific tasks, such as uploading meter results to a secure website and displaying reports.
  Other Names: DIDGET World Web Community

SUMMARY:
The purpose of this study is to evaluate a Diabetes data management program in the hands of potential users, both lay persons and healthcare professionals. With this data management system glucose results from the DIDGET TM meter can be uploaded to a secure website and used by adults with diabetes, by parents and guardians of children with diabetes, and by health care professionals to monitor diabetes by recognizing trends and patterns in blood sugar levels.

DETAILED DESCRIPTION:
Diabetes data management programs upload glucose meter results to computers to provide information to lay persons and their health care professionals. With this data management system glucose results from the DIDGET TM meter can be uploaded to a secure website and used by adults with diabetes, by parents and guardians of children with diabetes, and by health care professionals to monitor diabetes by recognizing trends and patterns in blood sugar levels. During the study subjects performed specific tasks, such as uploading meter results and displaying reports. The study evaluates the subjects' success in using the software program, the program's ease of use, clarity and usefulness of user instructions, and user satisfaction with the diabetes data management program.

ELIGIBILITY:
Inclusion Criteria:

* Lay users must be:

  1. Be at least 18 years of age
  2. Have diabetes or be the parent or legal guardian of a child with diabetes
  3. Be testing blood sugar at home at least twice daily for at least one month or be the parent or legal guardian of a child who has been testing blood sugar at home at least twice daily for at least one month
  4. Be able to speak, read, and understand English
  5. Have experience using a PC, navigating software programs, or browsing the internet
* Healthcare professionals must:

  1. Have experience using the internet
  2. Have experience using diabetes data management software in the medical office

Exclusion Criteria:

1. Person working for a competitive medical device company
2. Person having a cognitive disorder or condition which, in the opinion of the investigator, would put the person at risk or compromise the integrity of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (1):
- AMCR Institute, Escondido, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended Users of the Software: 35 young adults (age 18 to 24) with diabetes, 12 Parents/legal guardians of children with diabetes, and 3 healthcare professionals who work with this population used a diabetes data management program.
Period: Overall Study
Arm/Group | Intended Users of the Software
Started | 51
Completed | 50 (One subject did not meet inclusion criteria; the data was not used in analysis.)
Not Completed | 1
Not completed — Did not meet inclusion criteria | 1

BASELINE CHARACTERISTICS:
Groups:
- Intended Users of the Software: Baseline measures were analyzed using only data for the young adults (18-24 years of age) and parents/guardians (18 to 47 years of age) of children with diabetes, not healthcare professionals. Data was not used from one subject withdrawn from the study because the subject did not meet inclusion criteria.
Arm/Group | Intended Users of the Software
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] — Baseline participants included young adults with diabetes (age 18 to 24)and parents/guardians (age 18 to 47) of children with diabetes; note healthcare professionals were not included in this measure. One young adult subject was withdrawn from the study (did not meet inclusion criteria) and the data was not used in the analysis.
  years | 26.9 [18 to 47]
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline measures were analyzed using only data for the young adults (18-24 years of age) and parents/guardians (18 to 47 years of age) of children with diabetes, not healthcare professionals. Data was not used from one subject withdrawn from the study because the subject did not meet inclusion criteria.
  Participants
    Female | 29
    Male | 18
Region of Enrollment [Number; unit: participants] — Baseline measures were analyzed using only data for the young adults (18-24 years of age) and parents/guardians (18 to 47 years of age) of children with diabetes, not healthcare professionals. Data was not used from one subject withdrawn from the study because the subject did not meet inclusion criteria.
  participants
    United States | 47

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Who Rated Ease of Performing Specific Tasks as Very Simple to Neither Simple Nor Difficult (<=3 Rating)
Description: Subjects rated ease of using the software with respect to specific tasks. The rating scale was:
  1. = Very Simple
  2. = Simple
  3. = Neither Simple nor Difficult
  4. = Difficult
  5. = Very Difficult
Time Frame: 1-2 hours
Population: One subject was withdrawn from the study and the data was not used in the analysis. The subject did not meet inclusion criteria.
Measure: Number; unit: participants
Arm/Group | Intended Users of the Software
Number analyzed (Participants) | 50
participants
  Log in to DIDGET World Reports | 50
  Upload DIDGET Meter | 50
  Accept DIDGET meter settings | 50
  Display Blood Sugar Trend Report | 50
  Display the Standard Day Report | 50
  Change Daily Time Periods | 40
  Display the Logbook | 49
  Display the Standard Week Report | 50
  Identify Out of Target Results | 50
  Print the Standard Day and Standard Week Reports | 50
  Display the Summary Report | 50
  Save Summary Reports as a file on your computer | 48
  Change Low and High Blood Sugar Ranges in Reports | 49
  Log out of Web Reports | 49

2. Secondary Outcome: Number of Participants Who Rated Clarity and Usefulness of User Instructions as Good to Excellent (>=3)
Description: After the software evaluation, subjects were asked to review the online help and rate it on a 5 point scale.
  1. = Unacceptable
  2. = Poor
  3. = Good
  4. = Very Good
  5. = Excellent
Time Frame: 1-2 hours
Measure: Number; unit: participants
Arm/Group | Intended Users of the Software
Number analyzed (Participants) | 50
participants
  Clarity of online help | 49
  Usefulness of online help | 47

3. Secondary Outcome: Number of Participants Who Rated Their Satisfaction With The Following as Good to Excellent (>=3)
Description: Subjects responded to questionnaires in rating features and appearance, usefulness, and satisfaction on a 5 point scale:
  1. = Unacceptable
  2. = Poor
  3. = Good
  4. = Very Good
  5. = Excellent
Time Frame: 1-2 hours
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intended Users of the Software
Number analyzed (Participants) | 50
participants
  Ease of getting started | 50
  Readability of computer display | 49
  Usefulness of Log Book Report | 50
  Usefulness of Blood Sugar Trend Graph | 50
  Usefulness of Standard Day Graph | 50
  Usefulness of Standard Week Graph | 50
  Usefulness of Summary Either Bar Or Pie Chart | 50
  Overall, type of information software gives me is | 50
  Overall, the ease of use of DIDGET World Reports | 49

4. Primary Outcome: Number of Participants Who Rated Successful (<=3) by Healthcare Professionals When Participants Performed Specific Software Tasks
Description: Study staff rated participants on their success at performing specific tasks. The rating scale was:
  1. = Successful ( no assistance)
  2. = Successful after staff prompted to view user instructions
  3. = Successful with verbal assistance or review of part of user instructions (as review a specific function during a Customer Service call)
  4. = Unsuccessful (Subject could not perform the task)
  5. = Subject could not perform task due to software or hardware failure after repeated attempt.
Time Frame: 1-2 hours
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intended Users of the Software
Number analyzed (Participants) | 50
participants
  Log in to DIDGET World Reports | 50
  Upload DIDGET Meter | 50
  Accept DIDGET meter settings | 50
  Display Blood Sugar Trend Report | 50
  Display the Standard Day Report | 50
  Change Daily Time Periods | 49
  Display the Logbook | 50
  Display the Standard Week Report | 50
  Identify Out of Target Results | 50
  Print the Standard Day and Standard Week Reports | 50
  Display the Summary Report | 50
  Save Summary Reports as a file on your computer | 50
  Change Low and High Blood Sugar Ranges in Reports | 50
  Log out of Web Reports | 48

ADVERSE EVENTS:
Arm/Group | Intended Users of the Software
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less